CLINICAL TRIAL: NCT06181513
Title: Effect of Probiotics on Cognitive Functioning of Patients With Mild Alzheimer's Disease
Brief Title: Probiotics in Mild Alzheimer's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Nicosia (Other)
Collaborators: Cyprus Institute of Neurology and Genetics (Other)
Responsible Party: Principal Investigator, Nicoletta Nicolaou, Associate Professor, University of Nicosia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AARG-NTF-22-928616
Record Dates: First submitted 2023-12-08; First posted 2023-12-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Neurodegenerative Diseases; Cognition Disorders in Old Age
Keywords: probiotics; Electroencephalogram (EEG); cognitive function; Alzheimer's Disease; neuropsychological testing; Electrocardiogram (EKG)
MeSH Terms: conditions — Neurodegenerative Diseases; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): Participants received 1 capsule daily of probiotics, administered orally for 16 weeks.
  Interventions: Drug: Probiotic Blend Capsule
- Placebo (Placebo Comparator): Participants received 1 capsule daily of placebo, administered orally for 16 weeks.
  Interventions: Drug: Probiotic Blend Capsule

INTERVENTIONS:
Drug: Probiotic Blend Capsule — 20 million CFU (Lactobacillus paracasei, Lactobacillus plantarum, Lactobacillus rhamnosus, Lactobacillus helveticus, Bifidobacterium breve)
  Other Names: Ultrabiotique Equilibre 30 Vitavea

SUMMARY:
The main objective is to investigate whether administration of probiotics to patients with mild Alzheimer's Disease (AD) reduces neuroinflammation, improves cognitive function and modifies neurophysiological measures, compared to a patient group that receives placebo (no active probiotics).

DETAILED DESCRIPTION:
We will measure specific blood inflammatory markers (primary outcome), neurophysiological activity, cognitive test scores, microbiome composition and dietary habits of participants in the probiotics and placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥65 years, able to give consent
* Mini-Mental State Examination (MMSE) scores 19-23 (mild AD)
* approximately equal male:female ratio

Exclusion Criteria:

* Inability to give consent
* other neurological disease
* relevant psychiatric disorders (e.g. major depression)
* gastrointestinal/metabolic conditions
* history of alcohol/substance dependence
* use of systemic antibiotics in the previous 6 months
* corticosteroid use
* immune stimulating medications
* immunosuppressive agents
* probiotics consumption in the previous 6 months.
* immunosuppression
* structural heart disease
* neutropenia
* radiation
* active intestinal disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Level of inflammatory markers | Baseline (week 0), end of study (week 16)
  Peripheral inflammation markers implicated in the pathogenesis of mild-AD (pro-inflammatory cytokines: IL-6, IL-1β, CXCL2, NLRP3; anti-inflammatory cytokines: IL-10. Isolated from blood plasma.

SECONDARY OUTCOMES:
Cognitive function and neuropsychological scores | Baseline (week 0), end of study (week 16)
  Mini-Mental State Examination (MMSE)
Cognitive function and neuropsychological scores | Baseline (week 0), end of study (week 16)
  Montreal Cognitive Assessment (MoCA)
Cognitive function and neuropsychological scores | Baseline (week 0), end of study (week 16)
  Rey-Osterrieth complex figure test
Cognitive function and neuropsychological scores | Baseline (week 0), end of study (week 16)
  Wechsler Abbreviated Scale of Intelligence (WASI)
Neurophysiological activity changes | Baseline (week 0), end of study (week 16)
  Electroencephalogram (EEG) and electrocardiogram (EKG) measured at rest (eyes open, eyes closed).
Microbiome profile | Baseline (week 0)
  16S rDNA gene sequencing for bacterial identification, taxonomic profiling.

OTHER OUTCOMES:
Dietary habits | Baseline (week 0)
  Food Frequency Questionnaire (confounding)

CONTACTS AND LOCATIONS:
Locations (1):
- The Cyprus Institute of Neurology and Genetics, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided